CLINICAL TRIAL: NCT03956693
Title: HEADS: UP (Helping Ease Anxiety and Depression Following Stroke) Psychological Self-management Intervention: Non-randomised Pilot Study
Brief Title: Helping Ease Anxiety and Depression Following Stroke
Acronym: HEADS:UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: University of Stirling (Other); Edinburgh Napier University (Other); The Stroke Association, United Kingdom (Other); Yunus Centre for Social Business and Health (Unknown); University of Strathclyde (Other); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SA PPA 18\100011 (stage 1)
Record Dates: First submitted 2019-05-08; First posted 2019-05-21 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Stroke; CVA (Cerebrovascular Accident); Anxiety; Depression
Keywords: Stroke; CVA (cardiovascular accident); Anxiety; Depression; Mindfulness; Mindfulness Based Stress Reduction; Self-management
MeSH Terms: conditions — Stroke; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HEADS: UP (Experimental): HEADS: UP is group-based mindfulness intervention based on the original mindfulness based stress reduction course, but adapted for people affected by stroke.
  Interventions: Behavioral: HEADS: UP

INTERVENTIONS:
Behavioral: HEADS: UP — HEADS: UP comprises 9 x 2.5 hour mindfulness teaching sessions and a silent retreat in week 7. Course materials include accessible information packs and resources to complement class-based sessions.
  The first week of the 9-week course is an introductory class. The purpose of the introductory class is to give participants the opportunity to meet the trainers and to decide if they want to learn more about mindfulness. The introductory session also allows participants to meet other people on the course and to share their (stroke) stories.

SUMMARY:
The aim of this mixed methods research is to conduct feasibility pilot testing of an existing mindfulness intervention called HEADS: UP. The intervention is designed to help people affected by stroke self-manage symptoms of anxiety and depression.

DETAILED DESCRIPTION:
Mindfulness-based interventions are thought to help people affected by stroke (Lawrence et al., 2013). Helping Ease Anxiety and Depression (HEADS: UP) is an adapted mindfulness-based intervention for people affected by stroke (Lawrence, 2019). This study aligns with the feasibility/piloting stage of the Medical Research Council framework (Craig et al., 2008) and will optimise intervention delivery and study processes, ensuring all elements are working together, ready for testing at a later stage.

The aim of this mixed methods research is to conduct feasibility pilot testing of HEADS: UP to help people affected by stroke self-manage symptoms of anxiety and depression prior to Phase III testing in future work.

This stage is a non-randomised pilot study based in Glasgow, United Kingdom. The purpose of the pilot is to assess feasibility and acceptability of delivering HEADS: UP, and recruitment and questionnaire data collection processes; identify any additional HEADS: UP adaptions.

ELIGIBILITY:
Inclusion Criteria:

* Have had ≥1 stroke 3-60 months previously (reflects incidence of anxiety/depression)
* Interested in learning skills to help them cope with self-reported anxiety and/or depression
* Able to speak and understand conversational English
* Able to identify a family member/peer who would: like to take part, can speak and understand conversational English; not participating in another trial.

Exclusion Criteria:

* Prior MBSR attendance in the last three years (as this may confound results)
* Current participant in another trial
* Cannot follow a 2-stage command
* ≥28 on Behavioural Assessment of Dysexecutive Syndrome (BADS) scale; assesses the cognitive skills required to engage with group-based interventions (goo.gl/uumeFw)
* Hospital Anxiety and Depression Scale (HADS); screens for anxiety and depression; used extensively in Primary Care research (goo.gl/TtdDDW). A score of 8-10 suggests mood disorder; ≥11 indicates 'probable presence'. A total cut-off score of 11 achieves optimal balance between sensitivity and specificity, and will be used for family/peer participants who have not had a stroke. A lower cut-off score is recommended for stroke survivors i.e. 4 on each sub-scale.

NOTE: A current prescription for anxiolytics or antidepressants is not an exclusion criterion. If screening identifies a potential participant who requires GP referral, that individual may subsequently be prescribed medication; this is a feature of the pilot work. In a future trial, where participants are randomised to two arms and there is equal probability of people being on medication in each arm, it will not be an issue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Stroke Specific Quality of Life Scale (SS-QOL): change is being assessed | Weeks 0, 9, 21
  The Stroke Specific Quality of Life Scale (SS-QOL) is an outcome measure intended to assess of health-related quality of life for people affected by stroke. It is a self-report scale containing 49 items in 12 domains. Items are rated on a 5-point Likert scale and the questionnaire is usually completed in 10-15 minutes.
Stroke Impact Scale (SIS): change is being assessed | Weeks 0, 9, 21
  The Stroke Impact Scale (SIS) is a self-report, health status measure for people affected by stroke. It was designed to assess strength, hand function, activities of daily living, mobility, communication, emotion, memory and thinking, and participation. The SIS can be used both in clinical and research settings. It contains 59 items and assesses 8 domains. Each item is rated using a 5-point Likert scale. A final single-item question assesses the individual's perception of recovery from stroke, measured using a visual analogue scale, where 0 = no recovery & 100 = full recovery. The scale is normally completed in 15-20 minutes.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS): change is being assessed | Weeks 0, 9, 21
  The Hospital Anxiety and Depression Scale (HADS) is a self-administered measure of depression and anxiety. The HADS is not a diagnostic tool, but can screen for anxiety and depression. The HADS has 14 items in total and asks about mood in the past week. Seven items assess depression and seven items assess anxiety. The HADS can be administered repeatedly without impacting on validity. Each item is rated on a 4-point scale and provide a score 0-21. A higher score indicates higher distress.
  Usually completed in 2-5 minutes
Depression Anxiety Stress Scale (DASS): change is being assessed | Weeks 0, 9, 21
  The DASS is a set of three self-report scales designed to measure depression, anxiety and stress. Each of the three DASS scales contains 14 items, divided into subscales of 2-5 items with similar content. The Depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest/involvement, anhedonia, and inertia. The Anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The Stress scale is sensitive to levels of chronic non-specific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset/agitated, irritable/over-reactive and impatient. Subjects are asked to use 4-point severity/frequency scales to rate the extent to which they have experienced each state over the past week. Scores for Depression, Anxiety and Stress are calculated by summing the scores for the relevant items.
Beck Depression Inventory II (BDI-II): change is being assessed | Weeks 0, 9, 21
  The Beck Depression Inventory 11 (BDI-II) is a 21 items self-report scale to assess the intensity of depression. Each item is a list of four statements arranged in increasing severity about a symptom of depression. Score range between 0-63 with higher score indicating greater severity.
  Normally completed in 5-10 minutes.
Beck Anxiety Inventory (BAI): change is being assessed | Weeks 0, 9 21
  The Beck Anxiety Inventory (BAI) is a self-report 21-item scale for measuring anxiety. The questions ask about symptoms of anxiety the subject has had during the past week. Each question is scored between 0 (mild) and 3 (severe) and a total score will vary between 0-63. Higher scores indicate more severe anxiety symptoms.
EQ-5D 5L: change is being assessed | Weeks 0, 9, 21
  The 5-level EQ-5D version (EQ-5D-5L) comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

OTHER OUTCOMES:
Carer Strain Index (CSI): change is being assessed | Weeks 0, 9, 21
  The Carer Strain Index (CSI) is a 13-item self-report questionnaire. The tool covers employment, financial, physical, social and time. Positive responses to 7 or more items on the index indicate a greater level of strain. This instrument can be used to assess individuals of any age who have assumed the role of carer for an older adult.
Focus Groups (FG): change is being assessed | Weeks 9, 21
  Focus Groups (FGs) will be used to collect qualitative data. Focus groups will explore the feasibility, acceptability, meaningfulness, and effectiveness of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Lawrence, PhD, Study Director — Glasgow Caledonian University
Locations (1):
- Glasgow Caledonian University, Glasgow, Glasgow (City Of), United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Lawrence, M. (2019) Helping Ease Anxiety and Depression After Stroke (HEADS: UP): Research Project Briefing from the Chief Scientific Office. Available at: www.cso.scot.nhs.uk (Accessed: 7 May 2019).
- [Background] Lawrence M, Booth J, Mercer S, Crawford E. A systematic review of the benefits of mindfulness-based interventions following transient ischemic attack and stroke. Int J Stroke. 2013 Aug;8(6):465-74. doi: 10.1111/ijs.12135. PMID 23879751
- See also: Helping Ease Anxiety and Depression after Stroke (HEADS: UP) - Research Briefing — https://www.cso.scot.nhs.uk/wp-content/uploads/HIPS1663RPB.pdf